CLINICAL TRIAL: NCT00595816
Title: Prevention of Musculoskeletal Injuries in Finnish Conscripts. A Cluster Randomized Controlled Trial.
Brief Title: Injury Prevention Among Conscripts
Acronym: VASTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UKK Institute (Other)
Collaborators: Finland's Slot Machine Association (RAY) (Unknown); Ministry of Education (Ambiguous); Scientific Advisory Board for Defence (MATINE) (Unknown)
Responsible Party: The Urho Kaleva Kekkonen Institute for Health Promotion Research, The UKK Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UKK VASTE
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Back Problems and Other Musculoskeletal Injuries
Keywords: low back pain; physical fitness; injury; prevention; conscripts
MeSH Terms: conditions — Low Back Pain; Wounds and Injuries | interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Active treatment: physical training and counselling
  Interventions: Other: physical training and counselling

INTERVENTIONS:
Other: physical training and counselling — Neuromuscular training program 3 times per week 30 minutes per session and counselling on back problems and other musculosceletal injuries

SUMMARY:
The purpose of this clinical trial is to study the effect of neuromuscular training program and regular safety counselling on the risk of musculoskeletal injuries in adolescent conscripts.

800 voluntary participants are recruited from the four army companies in western Finland during the years 2007 and 2008.

ELIGIBILITY:
Inclusion Criteria:

* healthy conscripts who gave informed consent for participation

Exclusion Criteria:

* disease or injury preventing physical training

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 800 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Musculoskeletal injuries | 12 months

SECONDARY OUTCOMES:
Intensity of low back pain, Physical fitness | 1,2,6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jari P Parkkari, MD, PhD, Principal Investigator — The UKK Institute
Locations (2):
- Finland (2):
  - Jari Parkkari, Tampere, P.O Box 30
  - Jari Parkkari, Tampere, Pirkanmaa

REFERENCES:
- [Background] Suni J, Rinne M, Natri A, Statistisian MP, Parkkari J, Alaranta H. Control of the lumbar neutral zone decreases low back pain and improves self-evaluated work ability: a 12-month randomized controlled study. Spine (Phila Pa 1976). 2006 Aug 15;31(18):E611-20. doi: 10.1097/01.brs.0000231701.76452.05. PMID 16915076
- [Derived] Suni JH, Taanila H, Mattila VM, Ohrankammen O, Vuorinen P, Pihlajamaki H, Parkkari J. Neuromuscular exercise and counseling decrease absenteeism due to low back pain in young conscripts: a randomized, population-based primary prevention study. Spine (Phila Pa 1976). 2013 Mar 1;38(5):375-84. doi: 10.1097/BRS.0b013e318270a12d. PMID 22941095
- [Derived] Parkkari J, Taanila H, Suni J, Mattila VM, Ohrankammen O, Vuorinen P, Kannus P, Pihlajamaki H. Neuromuscular training with injury prevention counselling to decrease the risk of acute musculoskeletal injury in young men during military service: a population-based, randomised study. BMC Med. 2011 Apr 11;9:35. doi: 10.1186/1741-7015-9-35. PMID 21481230